CLINICAL TRIAL: NCT02601651
Title: Effect of Perioperative Intravenous Lidocaine on Opioid Consumption and Pain After Laparoscopic Totally Extraperitoneal Inguinal Hernioplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Anup Ghimire, Resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRC/520/015
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Pain, Postoperative
Keywords: Totally Extraperitoneal Inguinal Hernioplasty; Lidocaine infusion; Postoperative opioid consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Experimental): Lignocaine group (Group A) will receive an intravenous (IV) bolus 1.5 mg/kg at induction followed by continuous infusion of 2 mg/kg/hr until the tracheal extubation.
  Interventions: Drug: Lidocaine
- Normal saline (Placebo Comparator): Normal saline group (Group B) will receive an intravenous normal saline bolus at induction followed by continuous infusion of normal saline until the tracheal extubation
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — Lignocaine group will receive an intravenous (IV) bolus 1.5 mg/kg at induction followed by continuous infusion of 2 mg/kg/hr until the tracheal extubation.
  Other Names: Lignocaine; Loxicard
  Arms: Lidocaine
Drug: Normal saline — Normal saline group will receive an intravenous normal saline bolus at induction followed by continuous infusion of normal saline until the tracheal extubation
  Arms: Normal saline

SUMMARY:
The primary objectives of this study is to access the effect of perioperative lidocaine infusion on total morphine requirement during the first 24 h postoperatively in patients who underwent laparoscopic totally extraperitoneal inguinal hernioplasty.

DETAILED DESCRIPTION:
The use of intravenous lidocaine can be considered as a multimodal approach to pain relief. This method of analgesia has been associated with reductions in post-operative pain, analgesic consumption, nausea, vomiting and length of hospital stay in various surgeries (abdominal, spinal, thoracic surgery) including laparoscopic procedure .The primary reason for delayed patient recovery and longer hospital stays after surgery is postoperative pain and ileus .Opioids are the mainstay drug to treat pain in the postoperative period. However, nausea, vomiting, postoperative ileus and further delay in patient recovery will be exacerbated by opioid administration.

the higher inflammatory response is observed in the early postoperative phase following TEP surgery compared to the conventional shouldice repair. Therefore, laparoscopic repair of inguinal hernia should not be seen as less traumatic than the conventional approach.

Low-dose IV lidocaine (typically 1.5-3 mg/kg/h) is easy to administer, has well-established analgesic, anti-hyperalgesic, and anti-inflammatory effects, and excellent safety record . Because postoperative pain is to a large extent an inflammatory phenomenon, administration of systemic local anesthetics, which have inflammatory modulatory properties, could significantly reduce pain and therefore allow more rapid discharge. In addition, intravenous lidocaine is an effective modality for treating visceral pain.

Objectives

Primary : To access the effect of perioperative lidocaine infusion on total morphine requirement during the first 24 h postoperatively in patients who underwent laparoscopic TEP for inguinal hernioplasty

Secondary:

* Postoperative NRS Scores at rest and during movement (i.e. deep breathing, coughing) (at PACU, 2, 4, 6, 8, 12 and 24h)
* Time to first perception of pain in the postoperative period
* Incidence of post operative nausea and vomiting, shivering, and tinnitus during the first 24h
* Quality of Recovery based on QoR-40 questionnaire at 24 h of the surgery.
* Patient satisfaction at 24 h of the surgery.
* Incidence of Chronic pain after TEP Repair at 3 months.

RESEARCH HYPOTHESIS Perioperative intravenous lidocaine administration will not decrease opioid requirements and pain scores during the first 24 h after TEP for inguinal hernioplasty.

METHODOLOGY Written informed consent will be taken for the procedure from all the patients. A total of 64 male subjects of ASA PS I and II undergoing laparoscopic totally extraperitoneal inguinal hernia repair will be enrolled in the study. The study will be carried out according to the principles of the Declaration of Helsinki and following CONSORT guidelines.

After preoperative evaluation, all of the patients will be premedicated with oral diazepam (0.1-0.2 mg/kg; not exceeding > 10 mg) at the night before and 2 hour before surgery.In order to assess pain patients will be familiarized about the use of the Numeric Pain Rating Scale (NRS) (0-10 cm) where 0 is no pain and 10 is the worst imaginable excruciating pain. They will also be informed that they will be asked about the intensity of the pain using NRS score and the site of pain (incisional pain or groin pain) in the postoperative period.

During the study, both the patient and the investigator observing the outcome will be blinded about the assignment of patient group. In the preoperative holding area, the patients will be randomly assigned into any of two groups using computer generated random number. Details of group assignment and case number will be kept in a set of sealed opaque envelope. The anesthesia staff will open the envelope and prepare the intravenous solutions accordingly. The attending anesthesiologist who is unaware of the group allocated will follow the standard general anaesthesia protocol during the study.

In the operating room standard monitoring device will be attached to monitor and baseline heart rate, non-invasive blood pressure and oxygen saturation will be recorded. A peripheral vein will be cannulated for administration of IV fluid with 18 G cannula. Preoxygenation will be done with 100% oxygen for 3 min. Induction will be done with IV fentanyl 1.5 μg/kg, propofol 2-2.5 mg/kg till cessation of verbal response and tracheal intubation facilitated with vecuronium 0.1mg/kg IV.

At induction, lidocaine group (A group) patients will receive 1.5 mg/kg of lidocaine (Loxicard®, Neon pharmaceuticals, India) IV bolus followed by infusion of 2 mg/kg/h. The Normal Saline group (B group) will receive same volume IV bolus at induction followed by continuous infusion until the tracheal extubation.

Patients in both the group will receive preincisional infiltration in three trocar sites with 6 ml of 0.25% bupivacaine.

In all groups, anesthesia will be maintained with oxygen and isoflurane, adjusting the end-tidal concentration of isoflurane to maintain Mean Arterial Pressure(MAP) within 20% of baseline. IV fentanyl 0.5 μg/kg will be supplemented intraoperatively if MAP and heart rate increase by 20% from the baseline after ensuring adequate end tidal concentration of isoflurane ,muscle relaxation and targeted range of ETCO2. After observing curare notch in capnograph, supplemental vecuronium IV bolus doses will be given . Paracetamol 1 gm IV infusion will be started after induction and given over 15 min. Any episode of intraoperative hypotension (MAP lower than 65 mmHg) and bradycardia (heart rate < 50 bpm) will be treated with ephedrine 5 mg and atropine 0.4 mg IV respectively.

Standardized surgical procedure for the hernia as described for endoscopic TEP for inguinal hernia repair will be followed. Ketorolac 30 mg IV will be given at the end of surgery and continued at 8 h intervals postoperatively. On the completion of surgery, residual neuromuscular block will be reversed with neostigmine 0.05 mg/kg IV and glycopyrrolate 0.01 mg/kg IV. Following successful tracheal extubation, infusion of the lidocaine or saline will be stopped and the patient will be transferred to the postanesthesia care unit (PACU).

Postoperative Care and observation On arrival to the PACU, non-invasive blood pressure, heart rate, respiration, primary and secondary outcome variables will be monitored by the blinded investigator. Pain including its site will be assessed at rest and on deep breathing or coughing by NRS every 15 mins for the first 1 h and then at 2, 4, 6, 8, 12 and 24 h after surgery. If the NRS for pain is more than 3 at rest, morphine 1mg IV boluses will be administered, and repeated at the interval of 5 min until NRS is ≤ 3 for the first 24 h. Ondansetron 4 mg IV will be administered for persistent nausea (lasting >5 min) or vomiting.

In our institution, no step-down high dependency unit is available and patients will be transferred to the surgical ward after at least 2 h stay in the PACU.

Outcome parameters will be observed at PACU, 2, 4, 6, 8, 12 and 24 h after surgery.

Calculation of Sample Size

Sample size calculation was based on previous study with the use of intravenous lidocaine infusion for inguinal herniorrhaphy (Kang and Kim, 2011). Mean (SD) fentanyl consumption in the first 4-8 h between the lidocaine and placebo were 15.7 (6.3) and 21.4 (8.4) μg. Cohen d was used to calculate the effect size and was found to be 0.76.

Sample size was calculated using an online statistical calculator (G power® version 3.0.1). It was estimated that a sample size of 29 patients in each study group would achieve a power of 80% to detect an effect size of 0.76 in the primary outcome measure of opioid consumption, assuming a type I error of 0.05. Assuming 10% drop-outs during the study period, a total of 32 patients will taken for the study.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with American Society of Anaesthesiologists physical status (ASA PS) I and II of age 18 to 65 years
* Patients undergoing laparoscopic totally extraperitoneal repair for unilateral/bilateral inguinal hernia.

Exclusion Criteria:

* Refusal to give consent.
* ASA physical status III or more.
* Inability to comprehend pain assessment score or severe mental impairment
* Patient who weighed < 40 kg or >100 kg
* Severe underlying cardiac rhythm disorder
* Renal or hepatic disease
* Allergic to local anaesthetics
* Epilepsy
* Patients on regular analgesics or anti-arrhythmic drugs

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Total morphine requirement during the first 24 h postoperatively | 24h

SECONDARY OUTCOMES:
Pain at rest and with coughing or movement using the NRS scale | 24h
Time to first perception of pain | 24h
Incidence of postoperative nausea and vomiting (PONV) will be evaluated on a three-point ordinal scale. | 24h
  0 = none, 1 = nausea, 2 = vomiting
Sedation score using five point scale | 24h
  0=alert, 1=arouses to voice, 2=arouses with gentle tactile stimulation, 3 = arouses with vigorous tactile stimulation, 4 = lack of responsiveness
Time to first voiding. | 24h
Quality of Recovery based on QoR-40 questionnaire at 24 h of the surgery. | 24h
Patient satisfaction using Likert Satisfaction Scale at 24 h following surgery | 24h
  1-Highly satisfied, 2-Satisfied, 3-Neutral, 4-Not satisfied, 5-Strongly dissatisfied
Other side effects such as light headedness, tinnitus, perioral numbness, arrythmia and pruritus will be documented. | 24h
Incidence of Chronic pain after TEP Repair | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Asish Subedi, MD, Study Director — B.P. Koirala Institute of Health Sciences
Locations (1):
- BP Koirala institute of health sciences, Dharān, Sunsari, Nepal

REFERENCES:
- [Derived] Ghimire A, Subedi A, Bhattarai B, Sah BP. The effect of intraoperative lidocaine infusion on opioid consumption and pain after totally extraperitoneal laparoscopic inguinal hernioplasty: a randomized controlled trial. BMC Anesthesiol. 2020 Jun 3;20(1):137. doi: 10.1186/s12871-020-01054-2. PMID 32493276